CLINICAL TRIAL: NCT00960349
Title: A Phase I, Open-label, Non-randomized Study, to Assess the Safety and Tolerability of Cediranib (AZD2171) in Combination With Cisplatin Plus a Fluoropyrimidine (Capecitabine or S-1) in Japanese Patients With Previously Untreated Locally Advanced or Metastatic Unresectable Gastric Cancer
Brief Title: Study of Cediranib Plus Cisplatin Plus Capecitabine/S-1 in Japanese Gastric Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00066
Record Dates: First submitted 2009-08-11; First posted 2009-08-17 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Japanese; PhI; Safety and tolerability; Cediranib in combination with cisplatin plus a fluoropyrimidine; Cediranib; Capecitabine; S-1; Cisplatin; Untreated locally advanced or metastatic unresectable gastric cancer (GC)
MeSH Terms: conditions — Stomach Neoplasms | interventions — cediranib; Cisplatin; S 1 (combination); titanium silicide; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Other): Cediranib 20mg + Cisplatin + S-1
  Interventions: Drug: Cediranib; Drug: Cisplatin; Drug: S-1
- Treatment B (Other): Cediranib 20mg + Cisplatin + Capecitabine
  Interventions: Drug: Cediranib; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Cediranib — Given orally at a dose of 20mg/day everyday until the patient meets any discontinuation criterion.
Drug: Cisplatin — Given as a intravenous infusion at a dose of 80mg/m2 over 2hours on Day 1 of each cycle followed by a 5-week rest period. A maximum of 8 cycles of cisplatin will be given.
  Other Names: Randa, Briplatin,
  Arms: Treatment A
Drug: S-1 — Given orally at a dose of 80 - 120mg/day according to BSA for 3 weeks followed by a 2-week rest period in each cycle. Will be continued indefinitely until the patient meets any discontinuation criterion.
  Other Names: TS-1
  Arms: Treatment A
Drug: Cisplatin — 60mg/m2 over 2hours on Day 1 of each cycle followed by a 5-week rest period. A maximum of 8 cycles of cisplatin will be given.
  Other Names: Randa, Briplatin
  Arms: Treatment B
Drug: Capecitabine — Given orally at a dose of 1000mg/m2 twice daily for 2 weeks followed by a 1-week rest period in each cycle. Will be continued indefinitely until the patient meets any discontinuation criterion.
  Other Names: Xeloda
  Arms: Treatment B

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of cediranib in combination with Cisplatin plus a Fluoropyrimidine (Capecitabine or S-1) in Japanese patients with previously untreated locally advanced or metastatic unresectable gastric cancer (GC).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of gastric adenocarcinoma (including the gastric cardia and esophagogastric junction)
* Having locally advanced or metastatic gastric cancer for which they must have received no prior systemic therapy for locally advanced disease. Previous gastrectomy, neoadjuvant and adjuvant therapy received > 6 months ago are acceptable
* Having a mild symptom in ordinal daily lives including walking and simple labour or works in the sitting position

Exclusion Criteria:

* A history of poorly controlled hypertension or resting BP > 150/100 mmHg in the presence or absence of a stable regimen of anti-hypertensive therapy or patients who are requiring maximal doses of calcium channel blockers to stabilize BP
* Significant Haemorrhage (> 30 ml bleeding/episode in previous 3 months) or haemoptysis (> 5 ml fresh blood in previous 4 weeks)
* Arterial thromboembolic event (including ischemic attack) in the previous 12 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety of each treatment arm will be measured in terms of adverse events, vital signs, clinical chemistry, haematology, urinalysis, electrocardiogram, and physical examinations. | Cycle 1 of each treatment arm

SECONDARY OUTCOMES:
Pharmacokinetics will be assessed in terms of Css,max, Css,min, tmax, AUCss and AUC0-8 for cediranib, and Cmax, tmax, AUC, AUC(0-t), CL or CL/F, t½λz for capecitabine, cisplatin and TS-1. Additional PK parameters may be determined. | Cycle 1 and 2 of each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Narikazu Boku, MD, Principal Investigator — Shizuoka Cancer Center, Japan
Locations (4):
- Japan (4):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Sayama, Osaka
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Chūō, Tokyo